CLINICAL TRIAL: NCT00106925
Title: Long-Term Evaluation and Follow Up Care of Patients Treated With Allogeneic Stem Cell Transplants
Brief Title: Long-term Evaluation and Follow-up Care of Patients Treated With Stem Cell Transplants
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050130; 05-H-0130
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-16

CONDITIONS: Graft-versus-leukemia; Graft vs Host Disease; Graft Rejection
Keywords: Peripheral Blood Stem Cells; Graft Versus Leukemia/Myeloma; Graft Versus Host Disease; Whole Body Irradiation; Leukemic Relapse; Natural History
MeSH Terms: conditions — Graft vs Host Disease; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: allogeneic stem cell transplant recipients
- 2: Donors

SUMMARY:
This study will provide follow-up evaluation and care of patients who have undergone allogeneic (donor) stem cell transplantation at the NIH Clinical Center. Patients are monitored for their response to treatment, disease relapse, and later-occurring effects of the transplant.

Patients between 10 and 80 years of age who received a donor stem cell transplant at the NIH Clinical Center under an NHLBI protocol may be eligible for this study. Candidates must have had their first transplant at least 3 years before entering the current study.

Participants are generally seen in the clinic every 12 months for some or all of the following procedures:

* Periodic physical examinations, eye examinations, and blood and urine tests.
* Bone marrow aspiration and biopsy: A sample of bone marrow is obtained for microscopic examination. The patient is given local anesthesia or conscious sedation. An area of the hipbone is numbed, a thin needle is inserted through the skin into the bone, and a small amount of marrow is withdrawn.
* Tissue biopsy: A small piece of tissue or tumor is obtained for microscopic examination. Depending on the site of the biopsy, the tissue may be removed using a cookie cutter-like "punch" instrument, a needle, or a knife. The area is numbed and the tissue is removed with the appropriate tool.
* Imaging tests to visualize organs, tissues, and cellular activity in specific tissues. For these tests, the patient lies on a table that slides into the scanner. They may include the following:

  1. Nuclear scans use a sensitive camera to track a small amount of radioactive material (radioisotope) that is given to the patient by mouth or through a vein. The scan may show abnormal areas of tissue in the bones, liver, spleen, kidney, brain, thyroid, or spine.
  2. Magnetic resonance imaging (MRI) uses a magnetic field and radio waves to examine small sections of body organs and tissues.
  3. Computerized tomography (CT) uses x-rays and can be done from different angles to provide a 3-dimensional view of tissues and organs.
  4. Positron emission tomography (PET) uses a fluid with a radioisotope attached to it to show cellular activity in specific tissues. The fluid is given through a vein and travels to the cells that are most active (like cancer cells), showing if there is an actively growing tumor.
* Pulmonary (lung) function tests: The patient breathes into a machine that measures the volume of air the person can move into and out of the lungs.
* Heart function tests may include the following:

  1. Electrocardiogram (EKG) evaluates the electrical activity of the heart. Electrodes placed on the chest transmit information from the heart to a machine.
  2. Echocardiogram (Echo) is an ultrasound test that uses sound waves to create an image of the heart and examine the function of the heart chambers and valves.
  3. Multiple gated acquisition scan (MUGA) is a nuclear medicine test that uses a small amount of radioactive chemical injected into a vein. A special scanner creates an image of the heart for examining the beating motion of the muscle.

Disease relapse or progression, or transplant-related problems may be treated with standard medical, radiation, or surgical therapy, or patients may be offered experimental therapy.

DETAILED DESCRIPTION:
While patients surviving more than three years from SCT have a high probability of being cured of their underlying disease, they are still at risk from several categories of complications which could remain lifelong risks including late recurrence (or continued persistence) of original disease, late effects from transplant related GVHD, immune dysfunction, or consequences from the chemotherapy and/or radiation given during transplant conditioning.

Since these complications are iatrogenic, the long term follow-up of SCT patients is the ethical responsibility of the transplant team. In addition, collecting data on late occurring complications allows for prospective evaluation of the long term consequences of surviving a particular transplant treatment approach (i.e. total body irradiation versus chemotherapy conditioning, T cell depleted versus T cell replete transplants).

This protocol is designed to allow for long term evaluation, data collection, and when needed, standard medical care of patients (and when appropriate their stem cell donor) who have received allogeneic stem cell transplantation in NHLBI protocols. This may include patients with bone marrow failure states, cytopenias, hemoglobinopathies, metastatic solid tumors, or hematologic malignancies.

No investigational treatments will be administered on this protocol. Participation will not constitute a promise of long-term medical care at the NIH, nor will it provide for the evaluation and treatment of any non-transplant related medical problems. This protocol will provide access to NIH hematologists experienced in the care of post transplant patients who can help transplant patients and their local physician manage post transplant complications. In return, data collected from subjects and their donors (when applicable) will provide NIH researchers valuable information and/or laboratory samples for the purposes of better understanding the long term consequences of stem cell transplantation and identifying areas in need of future research.

ELIGIBILITY:
* INCLUSION CRITERIA-TRANSPLANT RECIPIENTS:

Patients surviving three years or more from date of first stem cell transplant who have been treated.

-With an experimental allogeneic stem cell transplant on a NHLBI HB protocol

Or

-With a standard of care allogeneic stem cell transplant on an NHLBI protocol

Or

-Selectively, when the allogenic transplant was conducted outside the NIH, but the subject has a special condition of interest to the research team

Age greater than or equal to 7 years old and age less than or equal to 80

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA-STEM CELL TRANSPLANT RECIPIENTS:

None, all patients meeting the inclusion criteria will be eligible

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and donors (when applicable) will be co accrued to this protocol once they have survived a minimum of three years from date of transplant.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2005-04-22 (Actual)

PRIMARY OUTCOMES:
Assure consistency of care over time for transplant patients such that outcome data can be meaningfully accrued. | Ongoing
  monitor late effects of treatment and provide or recommend appropriate management

SECONDARY OUTCOMES:
Monitor the late effects of treatment and provide or recommend appropriate management | ongoing
  To collect long-term follow-up data and laboratory research samples on SCT recipients to determine outcomes for particular transplant treatment approaches.
Describe natural history of the primary disease process. Provide fellowship training in Hematology and Oncology. | ongoing
  Patients will be evaluated at 4, 5 and 7 years post-transplant, then every 5 years after that to monitor the natural history of their disease, to evaluate the long term effects of transplantation, and to provide for or recommend appropriate clinical management

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Le RQ, Melenhorst JJ, Battiwalla M, Hill B, Memon S, Savani BN, Shenoy A, Hensel NF, Koklanaris EK, Keyvanfar K, Hakim FT, Douek DC, Barrett AJ. Evolution of the donor T-cell repertoire in recipients in the second decade after allogeneic stem cell transplantation. Blood. 2011 May 12;117(19):5250-6. doi: 10.1182/blood-2011-01-329706. Epub 2011 Mar 18. PMID 21421838
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2005-H-0130.html